CLINICAL TRIAL: NCT06056063
Title: Evaluation of Novel CT Imaging for Simulation on a Linear Accelerator
Brief Title: Project Looking-Glass Evaluation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPCC 02923; 852966 (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2023-08-28; First posted 2023-09-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cone-Beam Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Evaluate the Halcyon 4.0 obtained CBCT in comparison to a CT SIM for radiotherapy dose planning (Experimental): To evaluate the Halcyon 4.0 as a machine that will obtain CBCT that will be comparable to a CT simulator for radiotherapy treatment planning dose calculation. The novel CBCT images of subjects with malignancies from six disease sites obtained during the course of treatment for evaluation in place of the standard evaluation CBCT will be compared to their initial standard conventional CT simulation images used for treatment planning.
  Interventions: Device: Halcyon 4.0

INTERVENTIONS:
Device: Halcyon 4.0 — This Halcyon 4.0 is a new imaging hardware recently developed by Varian and approved by the FDA.

SUMMARY:
Pilot study to validate the new design and workflow of Cone-Beam CT imaging for radiation therapy treatment simulation.

DETAILED DESCRIPTION:
This study is a prospective, non-randomized imaging evaluation study. A cohort of subjects undergoing standard of care radiation therapy will be selected based on malignancies from six disease sites. The Halcyon 4.0 images acquired in place of standard evaluation CT scans during the course of treatment will be used for target volume delineation and normal structures segmentation. Treatment plans will be recalculated based on the Halcyon 4.0 images from this system and compared to the original treatment plan. Dose differences will be evaluated. Two-tailed t-test will be used to compare the statistical significance of the dosimetric results as well as the volumetric differences among target volume and the volumes of organs at risk.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be treated with external beam radiotherapy at the Perelman Center for Advanced Medicine for any of the following malignancies: head-and-neck, thoracic, breast, gastrointestinal, gynecologic, or genitourinary.
* Age ≥ 18 years
* Ability to understand the requirements of the study and to give written informed consent, as determined by the treating physician
* Availability of a complete set of treatment plans, including CT simulation images, target and normal structure contours, and radiation treatment prescriptions

Exclusion Criteria:

* Subjects who are pregnant or have plans for pregnancy during the period of treatment.
* Any malignancy not stated above.
* Those unable to be treated on any linear accelerator (whether Truebeam™ or Halcyon™) unit either due to subject anatomy or treatment plan.
* Those undergoing proton therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-11-19 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of image quality of the novel cone-beam CT imaging system compared to that of standard cone-beam CT imaging and that of conventional fan beam CT imaging used for radiotherapy planning purposes | 1 year
  Qualitative results (Yes is acceptable/No is not acceptable) will be reported as tabulated data to demonstrate the differences from the standard practice
Ease of use of the novel cone-beam CT imaging system compared to standard practice | 1 year
  Ease of use of the novel cone-beam CT imaging system on a scale of 1 (very easy to use, no difficulty) to 5 (unable to use due to difficulty)
Quantitative comparison of the image quality of the novel cone-beam CT imaging system to that of standard cone-beam CT imaging and that of conventional fan beam CT imaging used for radiotherapy planning purposes | 1 year
  A scale of Better/Worse/Equal will be used for metrics such as CBCT image artifact, CBCT image quality for OAR contouring, CBCT image quality for GTV contouring, motion artifacts, auto-segmentation ability, electron density similarity
Statistical significance of quantitative comparison of the image quality of the novel cone-beam CT imaging system and standard practice | 1 year
  For situations that the quantitative results will be measured, such as the structure volume or predicted electron densities etc., statistical significance will be calculated.

SECONDARY OUTCOMES:
Evaluation of the suitability and workflow of the novel CBCT images for radiation treatment planning and dose calculation. | 1 year
  The secondary endpoint is to compare the accuracies of dose and volume calculations to the standard arm using the conventional CT simulation.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Alonso-Basanta, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No